CLINICAL TRIAL: NCT04916938
Title: Post-natal Post-traumatic Stress: Impact of an Early Dyadic Intervention Though Interaction Guidance Therapy on Maternal Sensitivity and Reduction of Maternal Stress
Acronym: EVAGIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180615; ID-RCB Number (Other: 2020-A02576-33)
Record Dates: First submitted 2021-03-19; First posted 2021-06-08 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: Post-Natal Post-traumatic Stress Disorder (PN-PTSD); Interactive guidance therapy; Video feedback
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Guidance Therapy (Experimental): Mother child psychotherapy based on video-feedback interaction after a free play session. The therapy usually enhances parent sensibility to the child.
  Interventions: Behavioral: Interaction Guidance Therapy; Behavioral: Interview; Behavioral: Self-rated questionnaires
- Treatment as usual (Active Comparator): Mother child psychotherapeutic sessions without video feed back.
  Interventions: Behavioral: Mother's child psychotherapeutic session; Behavioral: Interview; Behavioral: Self-rated questionnaires

INTERVENTIONS:
Behavioral: Interaction Guidance Therapy — Mother child psychotherapy based on video-feedback interaction after a free play session. The therapy usually enhances parent sensibility to the child.
  Arms: Interactive Guidance Therapy
Behavioral: Mother's child psychotherapeutic session — Mother's representation of the event, mother's representation of the relation to her child, maternal emotions.
  Arms: Treatment as usual
Behavioral: Interview — History and perception of the mother's issues.
Behavioral: Self-rated questionnaires — Parental Self-Questionnaire to assess the perception of the evolution of the father, mother and child

SUMMARY:
The aim of this study is to assess if an early therapeutic management focused on the mother-baby interaction using Interaction Guidance Therapy (IGT) with video feedback, brings an improvement of the maternal sensitivity in the interaction but also a decrease of the post-traumatic maternal symptoms.

Post Natal Post traumatic stress is known as a disorder that impaired maternal mental health but also development of motherhood and the construction of the bond to the baby through interactive disturbances.

The investigators will screen, among women who had a traumatic perception of an event related to the pregnancy or the childbirth, those who still present posttraumatic stress symptoms at 4 weeks post-partum. Four weeks from the traumatic event is the minimum delay to qualify a PTSD.

After randomization IGT versus Treatment As Usual (TAU), the investigators planned an early therapeutic intervention, 3 sessions at 8, 10 and 12 weeks of post-partum.

The investigators will assess the effect of the IGT on Maternal sensitivity and on the intensity of post-traumatic stress symptoms at 3 month post-partum and 1year.

DETAILED DESCRIPTION:
The investigators will compare the efficacy of Interactive Guidance Therapy, a parent-infant psychotherapy using video feed back versus a dyadic treatment conduct as usual (TAU) in women who present a post traumatic stress disorder related to childbirth or pregnancy.

The main assessment is the maternal sensitivity, assessed during a video recorded free play interaction between the mother and the baby and rate with the Coding of interactive Behaviour (CIB).

This is a Single Blind Randomized clinical trial. Only the rating of the (CIB), which is the primary end point, will be done blind for the treatment the dyad received.

The randomization will proceed after the inclusion visit and the first assessment that take place at 6 weeks of post partum.

The following assessments will take place at 4 months and 12 months. The investigators will conduct a national multicentre study with 5 inclusions centres, which are all child psychiatry unit specialized in perinatal period and already train or in training for the IGT method.

* Pre-screening in post partum ward or during post partum consultation.
* Pre Inclusion at 5 (+-1) weeks to assess PTSD with Post traumatic checklist (PCL -5)
* Inclusion and First assessment at 6 weeks post partum
* Randomization: 3 session of IGT or TAU at 8 weeks, 10 weeks and 12 weeks Assessment at 4 months (+/-2W) and 12 months (+/- 1M)

ELIGIBILITY:
Inclusion Criteria:

For the mother:

1. Mother over 18 years old, who gave birth to a healthy child
2. Mother having a PCL-5 score higher than > 31, 5 +/- 1 week after delivery and the traumatic event is related to childbirth or pregnancy.
3. Mother Speaking and reading French,
4. Mother with signed consent
5. Mother with rights open to social security
6. Mother and Father consent to the participation of the baby

For the father:

1. holder of parental authority
2. Speaking and reading French
3. Consent to self-reported questionnaires

Exclusion Criteria

1. PTSD not related to pregnancy or birth.
2. Child's health situation who impact the feasibility of the protocol, with a risk of hospitalization of more than 3 days between 6 and 12 weeks of life
3. Childbirth under 34 weeks of gestational age
4. Twins
5. Stillbirth
6. Any mother's acute, somatic or psychiatric clinical condition not compatible with the research procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Maternal sensitivity | At 4 months
  Evaluate by Coding Interactive Behaviour (CIB)

SECONDARY OUTCOMES:
Maternal sensitivity at 12 months | At 12 months
  Evaluate by Coding Interactive Behaviour (CIB)
Prevalence of PN-PTSD | At 4 months
  Evaluate by Post-traumatic stress disorder Checklist version DSM-5 (PCL-5)
Prevalence of PN-PTSD | At 12 months
  Evaluate by Post-traumatic stress disorder Checklist version DSM-5 (PCL-5)
Prevalence of post natal depressive symptoms | At 4 months
  Evaluation by Edinburgh post natal depression scale (EPDS)
Prevalence of post natal depressive symptoms | At 12 months
  Evaluation by Edinburgh post natal depression scale (EPDS)
Infant development ASQ | At 12 months
  assessed with questionnaire fulfilled by both parents Age and Stage Questionnaire-12 (ASQ-12) Minimal score is 0 (worse) - Maximal score is >= 30
Infant symptoms SCL | At 12 months
  assessed with questionnaire fulfilled by both parents : Symptoms Checklist (SCL) Minimal score is 0 (worse) - Maximal score is >= 30
fathers' Post-traumatic stress disorder | At 4 months
  assessed with Post-traumatic stress disorder Checklist (PCL-5) Minimal score is 0 Maximal score is 80 (worse)
fathers' Post-traumatic stress disorder | At 12 months
  assessed with Post-traumatic stress disorder Checklist (PCL-5) Minimal score is 0 Maximal score is 80 (worse)
Father's depressive symptoms | At 4 months
  assessed with Edinburgh post natal depression scale (EPDS) Minimal score is 0 - Maximal score is 30 (worse)
Father's depressive symptoms | At 12 months
  assessed with Edinburgh post natal depression scale (EPDS) Minimal score is 0 - Maximal score is 30 (worse)
both parents' anxiety | At 4 months
  assessed with State Trait Anxiety Inventory (STAI) Minimal score is 20 - Maximal score is 80 (worse)
both parents' anxiety | At 12 months
  assessed with State Trait Anxiety Inventory (STAI) Minimal score is 20 - Maximal score is 80 (worse)
both parents' perception of social support | At 4 months
  assessed with Social Support Scale (SSQ) Minimal score is 0 (worse) - Maximal score is 54
both parents' perception of social support | At 12 months
  assessed with Social Support Scale (SSQ) Minimal score is 0 (worse) - Maximal score is 54
both parents' perception of their marital relationship | At 4 months
  assessed with Dyadic Adjustment Scale (DAS) Minimal score is 16 (worse) - Maximal score is 96
both parents' perception of their marital relationship | At 12 months
  assessed with Dyadic Adjustment Scale (DAS) Minimal score is 16 (worse) - Maximal score is 96
both parents' bonding to the child | At 4 months
  assessed with Post-partum Bonding questionnaire (PBQ). Minimal score is 0 - Maximal score is 125 (worse)
both parents' bonding to the child | At 12 months
  assessed with Post-partum Bonding questionnaire (PBQ). Minimal score is 0 - Maximal score is 125 (worse)

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère BEAUQUIER-MACCOTTA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (10):
- France (10):
  - CHU Besançon, Besançon
  - CHU - Maternité, Besançon
  - Centre hospitalier Intercommunal André Grégoire, Montreuil
  - Etablissement Ville Evrard, Noisy-le-Sec
  - Centre hospitalier Saint Anne, Paris
  - Hôpital Saint Joseph - Maternité, Paris
  - Hôpital Necker - Enfants malades - pedospychiatrie, Paris
  - Hôpital Necker - Maternity, Paris
  - CHRU Reims, Reims
  - Centre hospitalier - unité de périnalité, Reims

IPD SHARING:
Plan to Share IPD: No